CLINICAL TRIAL: NCT04187105
Title: BMT-06: Phase II Study of Intensity Modulated Total Marrow Irradiation (IM-TMI) in Addition to Fludarabine/Cyclophosphamide and Post-Transplant Cyclophosphamide Conditioning for Partially HLA Mismatched (Haploidentical) Allogeneic Transplantation in Patients With Acute Leukemia and Myelodysplastic Syndrome (MDS)
Brief Title: BMT-06: Study of Intensity Modulated Total Marrow Irradiation (IM-TMI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1149
Record Dates: First submitted 2019-11-11; First posted 2019-12-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia; MDS
Keywords: Stem Cell Transplant; Half-matched (haploidentical) stem cell transplant
MeSH Terms: interventions — Transplantation Conditioning; Stem Cell Transplantation; fludarabine; Cyclophosphamide; Whole-Body Irradiation; Mesna; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Single group assignment to Arm 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Conditioning regimen with half-matched (haploidentical) stem cell transplant (Other)
  Interventions: Radiation: Conditioning regimen with half-matched (haploidentical) stem cell transplant; Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant; Device: Conditioning regimen with half-matched (haploidentical) stem cell transplant; Other: Conditioning regimen with half-matched (haploidentical) stem cell transplant

INTERVENTIONS:
Radiation: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Experimental: Total marrow irradiation 1.5 Gray (Gy) twice a daily on days -3 and -2
  Other Names: Total Marrow Irradiation
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — All patients will receive the following standard conditioning regimen:
  Fludarabine 30 mg/m2 IVPB daily from Day -6 (6 days before stem cell infusion) through Day -2
  Other Names: Fludarabine
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Cyclophosphamide 14.5 mg/kg intravenously prior to transplant on Days -6 and -5
  Other Names: Cyclophosphamide
Device: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Total body irradiation 2Gy on Day -1.
  Other Names: Total body irradiation
Other: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Stem cell infusion on Day 0.
  Other Names: Stem cell transplant
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Mesna 14.5 mg/kg IV starting 30 minutes prior to cyclophosphamide on Days -6 and -5 and continuing for at least 12 hours after end of cyclophosphamide
  Other Names: Mesna
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Cyclophosphamide 50 mg/kg IV on Days 3 and 4 after transplant at a dose of 50mg/kg per day
  Other Names: Cyclophosphamide
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Mesna 10 mg/kg IV every 4 hours for 10 doses starting 1 hour prior to cyclophosphamide on Days 3 and 4
  Other Names: Mesna
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Tacrolimus 0.03 mg/kg IBW Q24H starting on Day 5
  Other Names: Tacrolimus
Drug: Conditioning regimen with half-matched (haploidentical) stem cell transplant — Mycophenolate mofetil (MMF) 15 mg/kg PO TID (maximum daily dose of 3g/day) starting on Day 5
  Other Names: Mycophenolate mofetil

SUMMARY:
This study is being done to see if the addition of a targeted form of radiation to standard conditioning regimen will increase the amount of cancer cells that are killed off in the bone marrow and reduce the chances that your disease may return. This description is called Intensity Modulated Total Marrow Irradiation (IM-TMI).

DETAILED DESCRIPTION:
This is a single arm phase II clinical trial. The usual conditioning regimen for haploidentical transplant is the use of chemotherapy (fludarabine/cyclophosphamide) before the transplant and further chemotherapy with cyclophosphamide after the transplant. In addition, a small dose of radiation is also given.

Patients will receive a standard conditioning regimen with fludarabine, cyclophosphamide and total body irradiation (Flu/Cy/TBI) prior to haploidentical hematopoietic stem cell transplant (HSCT). Graft-versus-host disease prophylaxis will include cyclophosphamide 50 mg/kg on Day +3 and 4 along with tacrolimus and mycophenolate mofetil.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18-75 years
2. Related donor who is, at minimum, Human Leukocyte Antigen (HLA) haploidentical. The donor and recipient must be identical at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. A minimum match of 5/10 is therefore required, and will be considered sufficient evidence that the donor and recipient share one HLA haplotype. In addition, unrelated donors who are mismatched at least one of the following loci: HLA-A, HLA-B, HLA-Cw, HLA-or DRB1.
3. Eligible diagnoses are listed below. Patient must have one of the following:

   1. Relapsed or refractory acute leukemia (including AML or ALL in CR2 and primary refractory leukemia).
   2. Poor-risk AML in first remission:

      * AML arising from MDS or a myeloproliferative disorder, or secondary AML
      * Poor risk molecular features including but not limited to presence of FLT3 internal tandem duplication mutation.
      * Poor-risk cytogenetics: Monosomal karyotype, complex karyotype (> 3 abnormalities), inv(3), t(3;3), t(6;9), MLL rearrangement with the exception of t(9;11), or abnormalities of chromosome 5 or 7
   3. Poor risk ALL in first remission:

      * Poor risk cytogenetics: Philadelphia Chromosome, t(4;11), KMT2A translocation, t(8;14), complex karyotype (⩾ 5 chromosomal abnormalities) and low hypodiploidy (30-39 chromosomes)/near triploidy (60-78 chromosomes)
      * Philadelphia-like ALL
      * Presentation WBC >30 × 109 for B-ALL or >100 109 for T-ALL
      * Age>35
      * Poor MRD clearance, defined as levels >1 × 10-3 after induction and levels >5 × 10-4 after early consolidation by flow cytometry
   4. Myelodysplastic syndromes (MDS) with at least one of the following poor-risk features:

      * i. Poor-risk cytogenetics (including but not limited to 7/7q minus or complex cytogenetics)
      * ii. IPSS score of INT-2 or greater
      * iii. Treatment-related or Secondary MDS
      * iv. MDS diagnosed before age 21 years
      * v. Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy
      * vi. Life-threatening cytopenias, including those generally requiring greater than weekly transfusions
      * vii. Poor risk molecular features including but not limited to the presence of BCOR, ASXL1, p53 or RUNX1 mutations
   5. Mixed lineage and biphenotypic leukemia
4. Adequate end-organ function as measured by:

   * a. Left ventricular ejection fraction ≥ 40%
   * b. Bilirubin ≤ 2.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST < 5 x ULN
   * c. FEV1 and FVC > 50% of predicted

Exclusion Criteria:

1. Presence of significant co morbidity as shown by:

   * a. Left ventricular ejection fraction < 40%
   * b. Bilirubin > 2.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST > 5 x ULN
   * c. FEV1 and FVC < 50% of predicted or DLCO <50% of predicted once corrected for anemia
   * d. Karnofsky score <70
   * e. History of cirrhosis
2. Patients unable to sign informed consent
3. Patient who have previously received radiation to >20% of bone marrow containing areas (assessed by radiation oncology physician)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of 1 year Graft-Versus-Host Disease (GVHD) free, relapse free survival (GRFS) survival | 1 year
  To evaluate the number of patients with acute leukemia or MDS who are GVHD-free, relapse free (GRFS) after 1 year of undergoing undergoing a treatment regimen of haploidentical stem cell transplant with conditioning and total marrow irradiation.

SECONDARY OUTCOMES:
The number of patients with greater than or equal to grade 4 non-hematologic toxicities | 1 year post-stem cell transplant
  Evaluate the incidence of greater than or equal to grade 4 non-hematologic toxicities
Engraftment rates | 30 days post-stem cell transplant
  Engraftment rates at Day 30
Rates of incidence of full donor chimerism | 30 days post-stem cell transplant
  Rates of incidence of full donor chimerism at Day 30
The rate of overall survival (OS) | 1 year post-stem cell transplant
  The rate of overall survival (OS)
The rate of event free-survival (EFS) | 1 year post-stem cell transplant
  The rate of event free-survival (EFS)
The rate of Grade II-IV and III-IV acute GVHD and limited/extensive chronic GVHD | 1 year post-stem cell transplant
  The rate of Grade II-IV and III-IV acute GVHD and limited/extensive chronic GVHD
The rate of progression at 1 year post transplant | 1 year post-stem cell transplant
  The rate of progression at 1 year post transplant
The rate of relapse at 1 year post transplant | 1 year post-stem cell transplant
  The rate of relapse at 1 year post transplant
The rate of non-morality (NRM) at 1 year post transplant | 1 year post-stem cell transplant
  The rate of non-morality (NRM) at 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Rondelli Damiano, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States